CLINICAL TRIAL: NCT06793891
Title: The Effectiveness of a Proprietary Ashwagandha Extract on Stress Reduction: A Three-Arm Randomized, Double-Blinded, Placebo Controlled Clinical Trial
Brief Title: Effects of Ashwagandha Extract on Stress Levels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Principal Investigator, Jessie Hawkins, PhD, Nutraceuticals Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 24-09-900
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Stress
Keywords: energy; fatigue; cognition; nutraceuticals; Ashwagandha
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plant Extract 1 (Experimental): Participants in this arm will take an ashwagandha root supplement each day for 60 days.
  Interventions: Dietary Supplement: ashwagandha root
- Plant Extract 2 (Experimental): Participants in this arm will take an ashwagandha root and leaf supplement each day for 60 days.
  Interventions: Dietary Supplement: ashwagandha root and leaf
- Placebo (Placebo Comparator): Participants in this arm will take an inert placebo each day for 60 days.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: ashwagandha root — This substance is extracted from the root of the plant.
  Arms: Plant Extract 1
Dietary Supplement: ashwagandha root and leaf — This substance is extracted from both the root and leaves of the plant.
  Arms: Plant Extract 2
Other: placebo — The inert placebo does not contain any of the plant matter.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of two proprietary ashwagandha extracts on stress levels, with secondary outcomes of cognition, energy, and sleep, as compared to a placebo.

DETAILED DESCRIPTION:
Participants will take one of two extracts or a placebo every day for 60 days; outcomes of stress, sleep, energy, and cognition will provide information on effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness and demonstrated ability to comply with all study procedures, as well as availability for the duration of the study
* Self reported high stress
* Baseline score of above-average stress levels on the NRI-SS
* Biological sex of woman; gender identification of female
* Aged 30 to 59, inclusive
* Good general health as evidenced by medical history and screening
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional month after the end of the study
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* Pregnancy, trying to conceive, or breastfeeding
* Currently smokes or vapes (i.e., tobacco, flavored items, marijuana, etc.) or has in the past year
* Consumes > 8 alcoholic beverages in an average week
* Is a primary caretaker for a child younger than 18 months of age
* Currently consumes an ashwagandha supplement or has consumed one regularly (defined as 1x week or more often) within the past 24 months
* Consumes any stress aid, medication, diet, or supplement intended to improve stress in any way
* Current or recent (within 60 days) history of taking thyroid medications, hypertensive drugs, CNS depressants, diabetic medications, benzodiazepines, or immunosuppressants
* Any liver or kidney disorder
* Known allergic reactions to any components of the intervention
* Positive COVID-19 test within 30 days of the study period
* Recent dramatic weight changes (10% change in body weight in the last 6 months)
* Introducing a new investigational drug or other intervention within 60 days before the start of the study
* Introducing a new lifestyle stress-reduction aid (i.e. physical activity, yoga, etc) within 60 days before the start of the study

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — biological sex of woman; gender identification of female
Enrollment: 60 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Post-test Cortisol Awakening Response, after controlling for baseline scores | 60 days
  salivary cortisol levels will be taken immediately after waking and 30 minutes later to produce a composite score
NRI-SS (Nutraceuticals Research Institute's Stress Scale) | 60 days
  This is a validated scale measuring 6 subdomains of stress. It is measured on a likert scale. Scores on each subdomain can range from 5 to 42, with higher scores indicating greater stress levels.

SECONDARY OUTCOMES:
NRI-ES (Nutraceuticals Research Institute's Energy Scale) | 60 days
  This is a validated scale measuring 6 subdomains of energy. It is measured on a likert scale. Scores on each subdomain can range from 5 to 42, with higher scores indicating greater energy levels.
NRI-Sleep (Nutraceuticals Research Institute's Sleep Scale) | 60 days
  This is a validated scale measuring 7 subdomains of sleep. It is measured on a likert scale. Scores on each subdomain can range from 5-42 with higher scores indicating greater quality of sleep
NRI-Cognition Scale | 60 days
  This is a validated scale measuring 6 subdomains of cognition. It is measured on a likert scale. Scores on each subdomain can range from 5-42 with higher scores indicating greater quality of cognitive health

CONTACTS AND LOCATIONS:
Locations (1):
- Nutraceuticals Research Institute, Huntsville, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Consent to share IPD will not been obtained from participants.